CLINICAL TRIAL: NCT01635842
Title: Informed Consent and Clinical Trials: a Survey on the Patient's Level of Understanding
Brief Title: Informed Consent and Clinical Trials
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: 11073; Informed Consent Project (Other Grant/Funding Number: 2011 Ethics Committee - AUSL of Bologna)
Record Dates: First submitted 2012-06-26; First posted 2012-07-10 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Informed Consent
Keywords: Patient; information leaflet; informed consent; awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To understand the patients' meaning of the informed consent process in clinical trials.

Objective of the study is:

* to assess, in a cohort of subjects included in clinical trials, whether the information and the informed Consent Forms conveyed to the patients have been understood
* to assess whether the choice to participate in a clinical trial is informed and aware

DETAILED DESCRIPTION:
Patient information and the Informed Consent Form (ICF) represent a focal point for an informed and aware participation in clinical research. As required by the Declaration of Helsinki no medical experimentation, including research on identifiable human material, can be undertaken without the subject has previously been informed about many issues, including goals, methods, anticipated benefits, possible risks and discomforts, commitment required and the possibility of withdrawing from the study at any time without explanation. All this information is essential to guarantee that the decision to enter a clinical trial is free, well informed and aware. Only when patients have collected and understood all the information needed, they are able to give their agreement to participate at the study and sign the ICF.

An interesting element that identifies a deficit of understanding is the so-called "therapeutic misconception". This term expresses the erroneous beliefs in which could incur a participant to a study, on the therapeutic value of the experimental therapy. Recent studies in the literature shows that a high percentage of patients agree to participate in order to derive a personal benefit. This view contrasts with the main objective of the clinical trial that has its own purpose just in obtaining new knowledge. While it is understandable that a person would expect a personal benefit is equally important that he would base his hopes on a solid rationale (i.e. expected benefits). Many other things, if not carefully understood, can lead to the "therapeutic misconception", including the concept of randomization, the risks related to the study, the time required to release his own informed consent, the reason for which has been asked to participate. Even the misunderstanding of just one of these elements may raise false hopes able to impact heavily on the final decision.

During the Ethical Committee meetings of the Azienda USL di Bologna (local health authority) all these points have been often discussed through the process of the RCT approval. For this reason the Ethical Committee decided to carry out a survey aimed to better understand the value and the meaning of ICF.

Initially, it has been conducted a literature review of studies, with particular attention to on those published from 2006 up to date. The common objective of these studies was to assess the understanding of the ICF by patients who were asked to participate in clinical trials (research Medline, keywords: informed consent, comprehension, clinical trials). These studies were in general survey conducted through interviews or questionnaires.

These studies have been conducted in cardiology, oncology, surgery, or treatment of pain. The studies were phase I, II, III or IV. In general, the results from these studies raise doubts on about the understanding of some important elements of the ICF. These doubts have emerged also from an Italian experience reported in on a thesis of Master's Degree in Economics and Management of Health Services. More in details, two studies have investigated the understanding of the informed consent, with particular attention to the issue of the "therapeutic misconception": in the study "Joffe", although 90% of participants were satisfied with the process of informed consent, many of them would not have been able to recognize non-standard cares of experimental treatments (74%), the potential additional risks related from the trial (69%), and the scientific uncertainty of the benefits of experimental therapy (70%). In the study "Bergenmar", even though 80% of the subjects feels that they have understood the important elements of the research, it seems that 65% do not recognize the experimental nature (not standard) of treatment, the 80% are not aware of the potential additional risks, and 75% are not aware about the fact that the experimental treatment is not scientifically proven to be the best treatment available. More significant factors emerged from the literature review, for example a high percentage of patients (67%) who did not live the process of informed consent as an important step to decide whether to participate to the trial. A study of 21 patients revealed that many had recognized as the main objective of the research the increasing of knowledge for the benefit of future patients, but only for a few of them this altruistic motivation was an important element in the final decision to participate.

The study promoted by the Ethical Committee of Azienda USL Bologna is observational, prospective and cross sectional. An ad hoc questionnaire has been developed on the basis of the literature available and through the discussion among Ethical Committee members, where also lay people are represented. The questionnaire has been discussed with the clinicians promoting clinical trials and tested with a group of patients enrolled in clinical trial. The self-administered questionnaire in 20 items long.

The questionnaire will be proposed to a cohort of subjects who have signed the ICF for a participation in an interventional clinical trial, not earlyer than 30 days have passed since the ICF signature.

ELIGIBILITY:
Inclusion Criteria:

* subjects or legal representatives (care givers, parents) who have signed the IC during the last 30 days for participation in an interventional clinical trial
* release an authorization to be contacted by the Ethics Committee of AUSL Bologna.
* able to read Italian

Exclusion Criteria:

* subjects enrolled in observations studies
* not release of authorization to be contacted by the Ethics Committee

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects or legal representatives (care givers, parents) who have signed the ICF during the last 30 days for participation in an interventional clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Therapeutic misconception cases among participants | From the 31st to the 40th day since the ICF signature of the clinical trial
  The question N° 18 has 4 answers. The patients who will answer "yes, for sure" will be considered cases of "therapeutic misconception".
  The study is qualtative. The assessment needs a multidimensional evaluation through many primary outcomes.
Time required to release the informed consent signed | From the 31st to the 40th day since the ICF signature of the clinical trial
  The question N. 7 wants to verify the time passed between the release of information by the investigator and the signature of the informed consent (Less than 1 hour, more than 1 hour, more than 1 day, more than 1 week).
Understanding of the possibilities / alternatives to experimental therapy | From the 31st to the 40th day since the ICF signature of the clinical trial
  The questions N. 15 and N. 16 want to verify the awareness of possible alternatives to the experimental therapy.
Comprehension of the significance of the informed consent | From the 31st to the 40th day since the ICF signature of the clinical trial
  The question N. 11 want to verify the patient's awareness about the significance of the informed consent.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Mosconi, Biology, Principal Investigator — Ethics Committee AUSL of Bologna
Locations (1):
- Ethics Commitee AUSL of Bologna, Bologna, Bologna, Italy